CLINICAL TRIAL: NCT05892575
Title: The Effect of Urinary Incontinence Management Program in Obese Elderly on Quality of Life, 'Coping With Incontinence' and Loneliness
Brief Title: The Effect of Incontinence Program Applied to Obese Elderly on Quality of Life, Coping and Loneliness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Şeyma SOYANIT ERASLAN, research assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OndokuzMay
Record Dates: First submitted 2023-03-06; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Primary; Incontinence, Urge; Incontinence Stress; Aging
Keywords: Coping methods; obese elderly; urinary incontinence; loneliness; quality of life
MeSH Terms: conditions — Obesity; Urinary Incontinence, Urge; Urinary Incontinence, Stress; Urinary Incontinence | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental:educt (Experimental): Training on improving the quality of life, coping with incontinence and kegel exercises will be given to obese elderly people over 65 years of age with urinary incontinence in the experimental group.
  Face-to-face training will be given to the elderly in the experimental group for a total of 5 weeks, once a week day (60 minutes). In the 4th week, reminder messages will be started over the phone. The 4th week kegel exercise chart and nutrition list will be given. In the 5th week, kegel exercise dance will be watched. Sending reminder messages from the phone will continue for 3 months.
  Interventions: Behavioral: improving quality of life, coping with urinary incontinence and kegel exercise training
- active comparator, control group (No Intervention): The elderly in the control group will not be interfered with.

INTERVENTIONS:
Behavioral: improving quality of life, coping with urinary incontinence and kegel exercise training — Face-to-face training will be given to the elderly in the experimental group for a total of 5 weeks, once a week day (60 minutes). In the 4th week, reminder messages will be started over the phone. The 4th week kegel exercise chart and nutrition list will be given. In the 5th week, kegel exercise dance will be watched. Sending reminder messages from the phone will continue for 3 months.
  Arms: experimental:educt

SUMMARY:
The goal of this: It was planned in a single-blind randomized controlled pre-test-post-test experimental research design. The aim of this study is to determine the effect of urinary incontinence management program on quality of life, coping with incontinence and loneliness in obese elderly.

The main questions it aims to answer are:

Does the Urinary Incontinence Management Program prepared for the obese elderly affect the quality of life, coping with incontinence and loneliness levels of the elderly in the experimental and control groups? After the Urinary Incontinence Management Program prepared for the obese elderly, is there an increase in the incontinence quality of life of the obese elderly in the experimental group compared to the obese elderly in the control group? After the Urinary Incontinence Management Program prepared for the obese elderly, is there an increase in the level of coping with incontinence of the obese elderly in the experimental group compared to the obese elderly in the control group? After the Urinary Incontinence Management Program prepared for the obese elderly, is there a decrease in the loneliness levels of the obese elderly in the experimental group compared to the obese elderly in the control group? After the Urinary Incontinence Management Program prepared for the obese elderly, is there an increase in the incontinence quality of life, coping with incontinence and loneliness levels of the elderly in the experimental group after the intervention compared to the pre-intervention?

DETAILED DESCRIPTION:
Worldwide, there is a transition from a young population structure to an aging population structure, and life expectancy at birth is increasing. As the global growth of the elderly population will continue, we are moving towards an aging world.

According to the World Health Organization, it is estimated that the population aged 60 and over will reach 2 billion by 2050. With increasing age, changes occur in every system in the body. One of these systems is the urinary system.

UI suggests that it may be an early marker of the onset of frailty. In the elderly; UI is expressed as the 4th most disturbing disease after angina, difficulty in ambulation and psychiatric disorders. Among the UI subtypes, stress urinary incontinence and urge urinary incontinence are the most common and urge urinary incontinence is seen especially in the elderly.

UI occurs as a result of deterioration in pelvic floor structure functions.Obesity is the best known and potentially the most modifiable risk factor for the development of UI, leading to pelvic floor deficiencies. There is a strong and positive relationship between obesity and urinary incontinence.

Compared with patients of normal weight, obese patients are approximately twice as likely to present with urinary incontinence.

Individuals may experience physical and psychosocial limitations due to UI, and their quality of life may be adversely affected. As a result of this situation, anxiety, depression, deterioration in sexual life, decrease in physical activity, loss of self-confidence and social isolation problems can be seen. All these conditions are in themselves associated with poor quality of life.

Urinary incontinence is rarely reported, especially in older adults, as it is believed to be a natural consequence of aging and that there is no clear management approach or cure. Therefore, individuals with UI do not seek help from family members or healthcare providers for urinary incontinence symptoms for various reasons. However, despite experiencing urinary incontinence, people may not seek treatment for reasons such as ignorance, ignorance, not being able to find time to go to the doctor, thinking about urinary incontinence as normal, or rejecting or hiding incontinence. Individuals with urinary incontinence do not seek help and try to cope with this problem on their own.

UI that negatively affects psychological and social well-being and quality of life; Decreased self-confidence of the individual brings along problems such as living alone and escaping from society. Individuals sometimes reduce or avoid social contacts and activities to control UI. This leads to increased social isolation and feelings of loneliness.

It is stated that conservative treatment methods can be used in the first-line treatment of urinary incontinence. In the guidelines of the European Association of Urology, it is emphasized that conservative treatment methods of urinary incontinence should be used as the first choice in the treatment of patients. Conservative treatment methods include lifestyle changes (weight loss, smoking cessation, diet regulation, regulation of fluid consumption), behavioral treatments, and pelvic floor muscle training. Among these methods, pelvic floor muscle exercises come to the fore. In the treatment of urinary incontinence of the frail elderly, pelvic floor exercises are included in the first-line treatment.

Incontinence is also related to nutrition. Nutrition can affect lower urinary system functions. In order to prevent or reduce UI, the European Urology Association 2020 guideline states that different lifestyle practices, such as reducing caffeinated beverages, regulating fluid intake, and quitting smoking, together with weight loss, have an effect on UI symptoms.

Some exercises can reduce urinary incontinence symptoms. Characterized by a gentle/gentle, slow and coordinated sequence of movements, Tai-Chi exercise is a suitable form of exercise for older adults as it involves minimal strain on the joints and cardiovascular system. Tai chi exercise is an easy-to-learn and ubiquitous exercise recommended for both men and women in conditions related to the pelvic area and for improving health in the elderly. In one study, Tai Chi improved the quality of life of elderly women with overactive bladder syndrome, emergency urinary incontinence. In another study, it was found that men with lower urinary tract symptoms performed tai chi and a significant result was obtained compared to men without lower urinary tract symptoms.

Health-promoting measures for older adults with UI are necessary to maintain their well-being and prolong healthy life expectancy. It will be important to create a training component/plan for this. Considering learning principles in planned adult education activities can contribute to the formation of an effective learning environment for adults. Knowles brought a different and systematic perspective to the subject of adult learning. In this context, training components can be prepared according to Knowles' adult learning principles.

It is recommended to use some models and theories, especially behavior modification theories, for those with incontinence problems to acquire healthy lifestyle behaviors. Health Belief Model (SIM) is one of the best models that can be used to develop knowledge, attitudes, beliefs about urinary incontinence and to create behavior towards kegel exercise, which is one of the effective methods in preventing urinary incontinence.

Studies for the prevention of urinary incontinence are limited in the literature, and interventional studies based on a theoretical background have not been found. In this study, the Incontinence Management Program based on Knowles' Adult Learning Principles and Health Belief Model will be used.

According to Knowles' Adult Learning Principles, which gives a different and systematic perspective to adult learning, no national or international study on obese elderly people has been found in the literature. At the same time, although SIM is used for more than one disease and various studies have been conducted, no study has been found to strengthen the motivation to change behavior in order to ensure continuity for obese elderly people. In addition, no study has been found in the literature in which the effectiveness of an education in which lifestyle behaviors based on Knowles' Adult Learning Principles and Health Belief Model, Kegel exercises and Tai Chi exercises are applied in the management of UI.

ELIGIBILITY:
Inclusion criteria:

* Standardized Mini Mental Test (SMMT) total score of 24 and above,
* 30 ≥ BMI ≥ 34.9 (obesity class 1) obese,
* 65 years and older,
* Those experiencing stress or urge urinary incontinence,
* Able to use smart mobile phone, use Whatsapp application,
* Those who do not have a health problem that prevents them from doing Kegel exercises.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria,
* Those with a history of incontinence surgery,
* Those who are morbidly obese,
* Having neurological and psychiatric disease,
* with pelvic organ prolapse,
* Having a disease affecting the genital and urinary system,
* those who cannot be communication.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incontinence Quality of Life - I-QOL Scale | Time Frame: 17 weeks
  The incontinence quality of life scale was developed by Wagner et al. in the USA in 1996 to determine the quality of life in patients with urinary incontinence. The validity and reliability of I-QOL in our country was done by Özerdoğan (2003). It has three sub-areas: limitation of behavior, psychosocial influence, and social isolation. In the Incontinence Quality of Life Scale (I-QOL), all items are evaluated on a five-point Likert-type scale as 1=a lot, 2=a lot, 3=moderate, 4=somewhat, 5=not at all. A maximum of 110 points can be obtained from the overall scale, 40 points from the behavior limitation sub-dimension, 45 points from the psychosocial impact sub-dimension, and 25 points from the social isolation sub-dimension. High scores indicate better quality of life than low scores.
Incontinence Awareness and Attitude Scale | Time Frame: 17 weeks
  The scale was developed by Avcı et al in 2017. The answers given to each statement in the scale are in the form of strongly agree, agree, undecided, disagree, strongly disagree, and the scale is in a 5-point Likert type. The scale does not have a total score. For the sub-dimension of coping with urinary incontinence, a minimum of 6 and a maximum of 30 are taken. In this study, only the coping with urinary incontinence sub-dimension of this scale will be used.
Urogenital distress inventory | Time Frame: 17 weeks
  The Turkish validity study of the urogenital distress inventory (UDI) was performed by Çam et al (2007).
  The scale is an inquiry form used to measure the presence of lower urinary tract symptoms and the degree of distress. UDI-6 consists of six questions and is graded on a four-point Likert scale. The first two questions are aimed at revealing irritative symptoms (urgency, frequency and pain), while the 3rd and 4th questions are aimed at stress symptoms, and the last two questions are for obstructive or voiding symptoms. Six questions ask about frequent urination, leakage due to a sense of urgency, leakage related to activity, coughing or sneezing, a small amount of leakage, difficulty in emptying the bladder, and pain or discomfort in the lower abdomen or genital area.
Health Belief Scale for Urinary Incontinence and Kegel Exercise: | Time Frame: 17 weeks
  The scale was developed by Avcı and Yıldırım (2019) based on the health belief model to determine individuals' beliefs about urinary incontinence and kegel exercises. The scale consists of 49 questions in 5-point Likert type and 6 sub-dimensions. The scale does not have a total score. In this study, this scale; Kegel exercise perception of benefit sub-dimension, kegel exercise disability perception sub-dimension and self-efficacy sub-dimension will be used. The scores obtained from the sub-dimensions and sub-dimensions of the scale are as follows: between 7-35 points for the perception of benefit sub-dimension of kegel exercise; Kegel exercise varies between 9-45 points for the perception of disability sub-dimension and between 5-25 points for the self-efficacy sub-dimension.
  Higher scores indicate that benefits are perceived as high for the perception of benefit, and obstacles are perceived as high for the perception of obstacles.
Loneliness Scale for the Elderly: | Time Frame: 17 weeks
  The scale was developed by de Jong Gierveld and Kamphuis in 1985 and revised by de Jong Gierveld and van Tilburg in 1999. The Turkish validity-reliability study of the scale was carried out by Akgül and Yeşilyaprak (2015). The scale, which has 11 questions in total, consists of 2 sub-dimensions. 6 items (2,3,5,6,9,10) of the scale consist of negative statements measuring emotional loneliness, and 5 items (1,4,7,8,11) consist of positive statements that measure social loneliness. The extent to which the situation contained in each statement in the scale is experienced by the person is determined by a 3-point Likert type rating. The rating is 0= yes, 1= maybe, 2= no. The lowest score on the scale is 0, and the highest score is 22. Total loneliness can be divided into four levels: Level 1; not alone / does not feel lonely (score 0-4); Level 2; acceptable loneliness (5-14 points); Level 3; very lonely (15-18 points); Level 4; It is very intense loneliness (score 19-22).

SECONDARY OUTCOMES:
Body Mass İndex Measurement (Weıght and Heıght) (Time Frame: 17 Weeks) | 17 weeks
  Body Mass Index Measurements Will Be Made Before and After The İntervention.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydın Avci, professor, Study Director — Ondokuz Mayıs University
Locations (1):
- Sinop Family Health Center No. 1, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The impact of pelvic floor muscle training on the quality of life of women with urinary incontinence: a systematic literature review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5962309/